CLINICAL TRIAL: NCT03929835
Title: A Phase Ⅱ, Randomized, Double-blind, Placebo-controlled Study to Investigate the Efficacy and Safety of Cannabis Oil for the Treatment of Subjects With Hidradenitis Suppurativa
Brief Title: Study to Investigate the Efficacy and Safety of Cannabis Oil for the Treatment of Subjects With Hidradenitis Suppurativa
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: withdrawn due to COVID-19
Sponsor: TO Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TO_HS01_2017
Record Dates: First submitted 2019-04-24; First posted 2019-04-29 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Hidradenitis Suppurativa
Keywords: Cannabis
MeSH Terms: conditions — Hidradenitis Suppurativa; Marijuana Abuse | interventions — nabiximols; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Avidekel Oil (Experimental): The cannabis oil, sort T1/C20 CBD as categorized by the MOH guidelines will be made from Avidekel strain and olive oil extract. Avidekel oil contains Δ9-Tetra-Hydrocannabinol (Δ9-THC) and Cannabidiol (CBD) in a 1:20 ratio and at a concentration of 30% CBD and 1.5% Δ9-THC. Each Avidekel oil drop is approximately 0.04 ml in volume containing about 12 mg CBD and 0.6 mg Δ9-THC.
  Interventions: Drug: Cannabis oil
- Placebo (Placebo Comparator): Patients in the control group will receive placebo oil containing olive oil and Chlorophyll.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabis oil — T1/C20 CBD
  Other Names: Avidekel Oil
  Arms: Avidekel Oil
Drug: Placebo — Olive oil with chlorophyl
  Other Names: Olive oil with chlorophyl
  Arms: Placebo

SUMMARY:
Hidradenitis Suppurativa (HS), is a chronic skin disease, manifested as inflamed areas of hair follicles around apocrine sweat glands found in areas most commonly the axillae, inguinal and anogenital regions. Patients experience great deal of physical pain as well as profound psychological problems. HS patients may also be prone to health complications and diseases. Treatment to date is limited and consist mainly of antibiotic administration and novel biological drug with up to 40% efficiency. Recently it was shown that cannabinoids reduces the folliculo pilosebaceous activity, most likely due to activating arachnoiditis, lipostat , anti-proliferative and anti-inflammatory agents and reduce inflammation inducing cytokines.

DETAILED DESCRIPTION:
Forty participants will be recruited over two years. After determine eligibility by examining the study criteria for inclusion and exclusion, the patient will be asked to sign the informed consent form.

The YAKAR form of medical cannabis license application and a confidentiality waiver form will be sent to the YAKAR. The physician will explain to the patients that his/her participation in the trial can be terminated at any time and will explain the medical license conditions: It is absolutely forbidden to:

* Use cannabis in the presence of minors or in public
* Drive under the influence of cannabis
* The participant shall take measures to prevent the theft of cannabis and inform the Investigator and the YAKAR of an attempt to steal or lose of cannabis.

When the patient license arrives, the patient will be scheduled an appointment for the first visit of the trial at the hospital. Tikun-Olam will be informed and asked to supply the patient product on the visit day. The copy of the patient's license will be included into the trial source documents.

The participants will be randomly assigned in a 1:1 ratio to receive Avidekel oil or placebo oil. Patients will receive the oils as drops applied under the tongue 3 times a day.

The duration of study participation for each subject is expected to be 12 weeks (84 days), about 4 weeks from visit 0 until receiving the license and 8 weeks trial,of which, six weeks of dose titration. Over the course of twelve weeks, four visits will be conducted and there will be 3 telephone evaluations. During first visit screening and enrolment will be conducted. The second visit will take place four weeks later where patients will receive the oils and start the trial, followed by a phone call evaluation at day 5-7 after starting the treatment and at week 2±2 days. Than a visit approximately four weeks later, following another phone call evaluation at week 5±2 days from treatment beginning, F Last visit will be conducted at week 8±3 days. In each visit, the relevant variables will be collected (Please refer to Table 3. Schedule of events). At the end of the eight-week experiment, patients from the treatment and control groups will be given the option to use the Avidekel oil for a period of one year. First, all the patients will use the drug in the open label phase for 8 weeks, during this period 3 phone calls and 2 visits in the hospital will be conducted, using PI-NRS and HS-PGA score to evaluate treatment success. Patients who will have at least 1 point reduction on the HS-PGA score will be permitted to continue to the 1 year follow-up. During that period 2 visits, six months and one year, will be conducted and the relevant variables will be collected (see Table 3). All visits will take place at the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects >20.
* Subjects who are diagnosed with moderate to severe Hidradenitis Suppurativa for at least 12 months prior to screening.
* Written informed consent from participant.
* For women, consent to avoid pregnancy during the trial.
* Consent to avoid driving during the influence of cannabis

Exclusion Criteria:

* Patients receiving any of the following medications: Astemizole, Cisapride, Pimozide or Terfenadine.
* Patients with severe heart disease.
* Subjects suffering from Epilepsy.
* Subjects suffering from anxiety disorder.
* Subjects who had psychotic condition in the past OR suffering from psychosis.
* Schizophrenia OR family history of Schizophrenia OR any other mental disorder.
* Significant psychiatric inheritance in a first-degree family member, especially in patients under 30.
* Pregnancy or intention to become pregnant during the study period
* Subjects with any other condition, which in the judgment of the investigator would prevent the subject from completing the study.
* Subjects suffering from chronic pain that does not necessarily is an outcome of the HS (Fibromyalgia, slipped disc).
* Any condition that the Investigator believes would interfere with the intent of the study or would make participation not in the best interest of the patient.
* Patients suffering from alcohol and/or substance abuse
* Surgery within 30 days prior to screening or scheduled surgery during the study period.
* Current participation in another drug or device clinical trial, or participation in such a clinical trial
* Lack of cooperation until the end of the study period.
* Patients with medical cannabis license
* Patients suffering from kidney disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Clinical response | From Week 0 to Week 8
  1 point reduction in HS-PGA score in treatment vs. control at week 8

SECONDARY OUTCOMES:
Safety: Participants experiencing Adverse Events (AE's) or Serious Adverse Events (SAE's) | Week 3, Week 6, six months and 12 months
  Participants experiencing Adverse Events (AE's) or Serious Adverse Events (SAE's)
Efficacy: Hidradenitis suppurativa Severity Index (HSSI) | 6 weeks, six months and 12 months
  Hidradenitis suppurativa Severity Index (HSSI)
Clinical response | 6 weeks of treatment
  Hidradenitis Suppurativa Clinical Response (HiSCR)
Changes from baseline | From Week 0 to Week 6, six months and 12 months
  Dermatology Quality of Life Index (DLQI)
Efficacy on pain levels: VAS pain scale | From Week 0 to Week 8, 16 weeks, six months and 12 months
  VAS pain scale 11-point numerical pain rating scale

CONTACTS AND LOCATIONS:
Locations (1):
- Haemek Hospital, Afula, Israel

IPD SHARING:
Plan to Share IPD: Undecided